CLINICAL TRIAL: NCT04787120
Title: A France-based Study for Squid Liquid Embolic Agent for the Embolization of Abdominopelvic Arterial Bleeding Syndrome: SQUIDperi Study: A Non-interventional, Prospective, Single-arm, Multicenter Study
Brief Title: Squid Liquid Embolic Agent for the Embolization of Abdominopelvic Arterial Bleeding Syndrome (SQUIDperi Study)
Acronym: SQUIDperi
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LOFFROY BALT 2020-1
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Arterial Bleed; Abdominal; Embolism Arterial; Pelvic Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with arterial abdominopelvic bleeding: Arterial abdominopelvic bleeding or imminent risk of bleeding
  Interventions: Device: SQUIDperi

INTERVENTIONS:
Device: SQUIDperi — Liquid embolic delivery syringes and micro-catheter

SUMMARY:
Abdominopelvic bleeding can occur due to numerous causes including for the vast majority, trauma, surgery complications and tumors. Interventional radiologists often exclude arterial acute hemorrhage using cyanoacrylate or a liquid embolic agent, but few prospective results have been published to assess their efficacy and safety. The historic and most studied liquid embolic agent to date is Onyx. Results in the treatment of acute peripheral non-neurologic hemorrhage have been detailed in a meta-analysis published in 2015. This systematic review found 19 articles presenting 131 patient cases and 150 lesions treated with Onyx from 2005 to August 2014. There were 11 case series and 8 case reports but no prospective trial. The most common presenting symptoms were of gastrointestinal (GI) origin (n = 51). Rebleeding of the baseline lesion occurred in 7/131 patients. No deaths resulting from complications of the embolic procedure were reported. One patient died of persistent hemoptysis after treatment with Onyx. No deaths were directly attributable to the use of Onyx.

During a peripheral embolization procedure with available embolic agents other than SQUIDPERI, residual feedings or collateral vessels became gradually less visible to the operator due to the high radiopacity of the liquid. It was therefore essential to develop an embolization system with lower radiopacity, or with radiopacity that decreases over time. Additionally, depending on the angioarchitecture and flow characteristics, it is important to have an embolic agent with various viscosities. SQUIDPERI is a liquid embolic agent with various viscosities and radiopacities. It is indicated for the embolization of lesions in the peripheral vasculature but its use is poorly reported as of today.

The purpose of this prospective non interventional multicenter study is to evaluate the safety and efficacy of SQUIDPERI for the treatment of abdominopelvic arterial acute bleeding or imminent risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with an arterial abdominopelvic bleeding or imminent risk of bleeding, including visceral, muscular or GI territories, requiring embolization, along with angiographic abnormalities
* Patient for whom the use of SQUIDperi had been decided for an embolization
* Patient or authorized representative dully informed and having no objection to the clinical data collection and medical file access
* Patient > 18 years

Exclusion Criteria:

* Patient with severe live failure
* Patient participating in another interventional study
* Vulnerable patients including pregnant women
* Patient not eligible for treatment with liquid embolic agent
* Patients presenting contra-indications to SQUIDperi as describes in the Informations For Use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring an embolization for the treatment of abdominopelvic arterial bleeding or imminent risk of bleeding including visceral, muscular or digestive territories, along with angiographic abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of embolization success at one month | 1 month
  Defined as the absence of re-intervention for re-bleeding from the target artery/arteries embolized during the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Loffroy R, Kobeiter H, Vidal V, Frandon J, Pellerin O, Dean C, Sammoud S, Vernhet-Kovacsik H, Derbel H, Aho-Glele LS, Chevallier O, Sapoval M. Ethylene-vinyl alcohol copolymer-based non-adhesive liquid embolic agent for transcatheter arterial embolization in patients with abdominal/pelvic arterial bleeding: A prospective, single-arm, multicenter cohort study. Diagn Interv Imaging. 2025 Jun;106(6):226-236. doi: 10.1016/j.diii.2025.02.001. Epub 2025 Feb 13. PMID 39952827